CLINICAL TRIAL: NCT06130852
Title: Training Workshops for Parents of Children With Attention Deficit Hyperactivity Disorder: Effects on the Child's Agitation. Preliminary Study.
Brief Title: Effects of Behavioral Training Groups for Parents of Children With Attention Deficit Hyperactivity Disorder
Acronym: PENDAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: RC31/20/0398; 2020-A02977-32 (Other: ID-RCB)
Record Dates: First submitted 2023-11-08; First posted 2023-11-14 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Deficit; Attention
Keywords: behavioral parent training
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Non-pharmacological treatments focusing on parenting skills are found in many recommendations.
  Programs for families of children with behavioral problems (attention deficit hyperactivity disorder, oppositional defiant disorder or conduct disorder) have been developed in several countries and adapted to ADHD. These programs take a similar approach: providing information about the disorder, changing in parents' view of their child's disorders, and didactic techniques that are known to be effective. These treatments enable parents to regain confidence in their parenting role, thanks to means of analysis (ABC model) and action (behavioral tools, such as reinforcement practice, token economy, time-out).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral Parent Training (Experimental): This program includes 10 thematic sessions aimed at changing the parent's view of their child by encouraging them to focus on appropriate behaviors. The sessions focus on specific themes such as positive attention, the principle of reinforcement, or even homework management.
  This program combines knowledge about ADHD with behavioral and cognitive techniques.
  Interventions: Behavioral: Behavioral Parent Training
- control group (No Intervention): no behavioral parent training

INTERVENTIONS:
Behavioral: Behavioral Parent Training — 10 thematic sessions aimed at changing the parent's view of their child by encouraging them to focus on appropriate behaviors. The sessions focus on specific themes such as positive attention, the principle of reinforcement, or even homework management.
  Arms: Behavioral Parent Training

SUMMARY:
The therapeutic care of Attention Deficit Hyperactivity Disorder (ADHD) children focuses on the child but also on his environment and in particular his family. This type of approach has long existed in Anglo-Saxon countries. This project aims to collect preliminary data to build study to valid efficacy of a parenting skills program for parents of ADHD children in France and on the child's hyperactivity.

DETAILED DESCRIPTION:
Attention deficit/hyperactivity disorder (ADHD) is a neurodevelopmental disorder affecting approximately 3-5% of an age group in France. Its manifestations affect individual in its everyday life. In 2014, the High Authority of the Health proposes recommendations for the children and the teenagers susceptible to present ADHD both for the screening and for the therapeutic. In this document, an important place is given to the family of these patients. Strong links are found between negative parental behaviours and a negative trajectory of ADHD symptomatology.

It seems essential to support and to guide these parents of children working in a different way, and for whom the specific educational approaches are known. Numerous counseling and parent training programs have been launched in the Anglo-Saxon countries since the 1980s. One of the most common methods is that proposed, which consists of a short therapy group, centered around a pedagogy on ADHD and its ecological consequences, as well as on the transmission of tools from behavioral theories aimed at reducing negative manifestations with the aim of improving relations between the ADHD children and his parents. This method come from a society different from ours and adaptation to French families is necessary. After several years of clinical experience in the care of ADHD children and their families, we developed a new program that draws heavily on the Barkley program for its beneficial effects, but combines the teaching of other recognized methods. We have been experimenting this program in current practice for 4 years at the CHU Toulouse at the rate of one session per year. At the moment, we only have family satisfaction evaluations. Nevertheless, the various Anglo-Saxon cognitive and behavioural programmes mentioned above show an overall improvement in the quality of life of families and in particular in the acceptance and management of everyday disorders.

The classically found effects are an improvement in the quality of life of families and in particular in the acceptance and management of disorders on a daily basis. Few or no effects are observed directly on the child using conventional assessment methods.

The main goal of this study is to collect preliminary data of the effects of the PENDAH Workshops on motor activity ADHD children.

ELIGIBILITY:
Inclusion Criteria:

* Parents of children with mixed ADHD or hyperactive/impulsive according to DSM5 criteria (children will arrive with a pre-established diagnosis, verified and validated by a team doctor)
* Children aged 7 to 11 years (± 6 months)
* Existence of a parental complaint or a request for specific help in managing the child's daily problems
* Parents who have agreed to participate in the PENDAH program
* No opposition from both parents
* French language spoken and understood by workshop participants

Exclusion Criteria:

* Parental conflict incompatible with obtaining the non-opposition of both parents
* For the child and based on the DSM-5 criteria:
* Gille de la Tourette syndrome
* A conduct disorder
* Autism spectrum disorder
* A suspected or proven intellectual deficit based on the child's medical assessments sent to the investigating doctor

Ages: 7 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Actual)
Dates: Start 2021-09-04 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-09-04 (Actual)

PRIMARY OUTCOMES:
Motor Activity | 5 months
  Accelerometer was calibrated at 30 Hz. Data were poached at 60 seconds. The variable used is the vector magnitude (VM), which accounts for accelerations of motion in the three planes of space and is expressed in counts/minute.
Motor Activity | 10 months
  Accelerometer was calibrated at 30 Hz. Data were poached at 60 seconds. The variable used is the vector magnitude (VM), which accounts for accelerations of motion in the three planes of space and is expressed in counts/minute.

CONTACTS AND LOCATIONS:
Overall Officials: Yves CHAIX, MD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- UHToulouse, Toulouse Cedex9, France

IPD SHARING:
Plan to Share IPD: No